CLINICAL TRIAL: NCT02738073
Title: Effects of Tranexamic Acid on Blood Loss and Transfusion Requirement Following Hip Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: 14RGOOD01
Record Dates: First submitted 2014-02-10; First posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Hip Fracture
MeSH Terms: conditions — Hip Fractures | interventions — Tranexamic Acid

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Drug: Control: Saline
- Interventional (Active Comparator)
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Control: Saline
  Arms: Control
Drug: Tranexamic Acid
  Arms: Interventional

SUMMARY:
Tranexamic acid (TA) inhibits fibrinolysis by binding to lysine binding-sites of plasminogen to fibrin. Fibrinolysis is stimulated by surgical trauma, and the administration of TA has been shown effective in decreasing blood loss both intra-operatively and in the immediate post-operative period in elective hip and knee arthroplasty patients. Both the timing and dosing of TA has been investigated in these patients. Subsequent blood transfusion rate has also been shown to decrease as result of TA administration. Despite the support for TA utilization that exists in the arthroplasty literature, the data is scarce regarding its administration during surgical treatment of hip fractures. This is patient population who is at high risk for transfusion due to symptomatic post-operative anemia. This study aims to investigate whether TA's advantageous effects in the arthroplasty patient population can be extrapolated to the more unstable, heterogeneous hip fracture patient population. If the study is able to show a difference in blood loss and transfusion requirement, the long term implications of this with regards to cost and mortality can be significant.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to Bryn Mawr Hospital with fracture of the femoral neck, intertrochanteric region, or subtrochanteric region of the femur will be considered for the study.

Exclusion Criteria:

Exclusion criteria include

* age under 18
* allergy to TA
* known current or history of venous thromboembolism (VTE)
* history of known coagulopathy or bleeding disorder
* current subarachnoid hemorrhage
* previous history of seizures
* current use of estrogen/progesterone therapy
* renal failure defined as creatinine clearance less than 30 ml/min4
* multiple fractures
* pregnant or breastfeeding women
* planned nonoperative management of the fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
calculation of blood loss during the perioperative period | participants will be followed for the duration of hospital stay, an expected average of 2-3 days
  This study aims to investigate the effect of tranexamic acid (TA) on blood loss and transfusion requirement during the perioperative period in patients who are admitted to the hospital with fracture of the hip and undergo surgical treatment. Both the drop in hemoglobin level from time of surgery (T0 being defined as just prior to surgery, while the patient waits in surgical holding area) over the subsequent several days, as well as post-operative transfusion rate, will be measured. The researchers' hypothesis is that both the hemoglobin drop and the subsequent transfusion requirement in patients who receive TA will be less than those who received saline placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- Bryn Mawr Hospital, Bryn Mawr, Pennsylvania, United States